CLINICAL TRIAL: NCT05190848
Title: Correlation of Microbiome and Metabonomics With IgA Nephropathy
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, XueQing Yu, professor, Guangdong Provincial People's Hospital
Other Study IDs: GDPH-IgAN-microbiome
Record Dates: First submitted 2021-12-27; First posted 2022-01-13 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: IgA Nephropathy
Keywords: IgAN microbiome metabolite
MeSH Terms: conditions — Glomerulonephritis, IGA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine、blood、Oral swabs、Pharyngeal swab、feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
IgAN is the most prevalent primary glomerulonephritis in China, is characterized by the deposition of IgA1 (particularly, galactose-deficient IgA1) in the glomerular mesangium. Galactosedeficient IgA1, supposed to be produced by Peyer patches in the mucosa-associated lymphoid tissue (MALT), is triggered by exposure to commensal or pathogenic bacteria, involved in the initial step in the pathogenesis of IgAN. Similar to intestinal flora, a disruption in oral flora is closely associated with the occurrence of many malignant tumors and autoimmune diseases. The relationship between oral and throat microflora and the occurrence of IgAN is unclear at present. The aim of the present study was to develop a preliminary model based on mucosa -specific microbes and clinical indicators to facilitate the early diagnosis of IgAN and obtain insights into its treatment.

DETAILED DESCRIPTION:
IgAN-microbiome is an investigator-initiated，multi-center，Observational study. This study will recruit IgA nephropathy patients who have not been treated with glucocorticoids and immunosuppressants for 6 months and have not taken antibiotics for 1 month and their family members. Feces, urine, blood, oral mucosal swabs, and pharyngeal swabs will be collected and tested for microflora and metabolites in these areas.

Similar samples from IgA nephropathy patients were collected after 2 months and 6 months, respectively, for bacterial community detection and metabolite detection, and the relationship between bacterial community change and metabolite change and disease progression was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* (1) Pathological changes of IgAN were confirmed by renal biopsy (2) Age ≥16 years (3) IgA deposition caused by secondary factors such as non-purpura glomerulonephritis, liver cirrhosis, SLE, HIV infection and hepatitis B virus associated nephritis (4) No antibiotics and/or functional foods (probiotics and/or prebiotics) for at least one month prior to sampling (5) No hormone or immunosuppressant treatment in the six months prior to sampling (6) No significant changes in diet or medication for at least one month (7) No other immune or autoimmune diseases, such as systemic lupus erythematosus (8) Signed informed consent

Exclusion Criteria:

1. Type I or type II diabetes
2. Pregnancy and menstrual period
3. Mental illness and inability to assess follow-up
4. Medically diagnosed intestinal diseases such as irritable bowel syndrome and inflammatory bowel disease
5. Viral hepatitis or other infectious diseases
6. One month before specimen collection, use laxatives including but not limited to polyethylene glycol electrolyte dispersant, enema and other laxatives

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: IgA nephropathy confirmed by renal biopsy and family members living with them
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with all-cause death | From trial initiation to any event first occurrence,the first to arrive will be evaluated up to 6 months
  Death for any reason.
Number of Participants with not meet the entry criteria | From trial initiation to any event first occurrence,the first to arrive will be evaluated up to 6 months
  not meet the entry criteria for any reason

CONTACTS AND LOCATIONS:
Overall Officials: Xueqing Yu, Study Chair — Guangdong Provincial People's Hospital; Xinling Liang, Study Director — Guangdong Provincial People's Hospital; Zhiming Ye, Study Director — Guangdong Provincial People's Hospital
Locations (5):
- China (5):
  - Sun Yat-sen Memorial Hospital Sun Yat-sen university, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guanzhou, Guangdong
  - The First Affiliated Hospital of Sun Yat-sen University, Guanzhou, Guangdong